CLINICAL TRIAL: NCT03519022
Title: Influence of Methylphenidate and Duloxetine Maintenance on Pharmacodynamic Effects of Cocaine
Brief Title: Behavioral Effects of Drugs: Inpatient (35)
Acronym: BED IN 35
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Craig Rush (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Craig Rush, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 43500
Record Dates: First submitted 2018-04-11; First posted 2018-05-08 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2018-07

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — Cocaine; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be maintained on oral placebo. Subjects will be maintained on placebo and methylphenidate during placebo maintenance. Cocaine will be administered acutely during placebo maintenance. Placebo will be administered acutely during placebo maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo oral capsule; Drug: Methylphenidate
- Duloxetine (Active Comparator): Subjects will be maintained on oral duloxetine. Subjects will be maintained on duloxetine and methylphenidate during placebo maintenance. Cocaine will be administered acutely during duloxetine maintenance. Placebo will be administered acutely during duloxetine maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo oral capsule; Drug: Methylphenidate

INTERVENTIONS:
Drug: Cocaine — The pharmacodynamic effects of cocaine will be determined during maintenance on placebo and duloxetine.
Drug: Placebo oral capsule — The pharmacodynamic effects of placebo will be determined during maintenance on placebo and duloxetine.
Drug: Methylphenidate — The pharmacodynamic effects of methylphenidate maintenance will be determined during maintenance on placebo and duloxetine.
  Other Names: Metadate®

SUMMARY:
This study will determine the influence of methylphenidate (Metadate®) and duloxetine (Cymbalta®), alone and in combination, on the reinforcing, subjective and physiological effects of cocaine.

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance abuse or dependence that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to cocaine, methylphenidate or duloxetine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Reinforcing Effects of Cocaine Following Placebo Maintenance. | Following at least 4 days of maintenance on placebo during inpatient admission.
  Number of cocaine doses earned by subjects on a progressive ratio schedule of reinforcement.
Reinforcing Effects of Cocaine Following Duloxetine Maintenance. | Following at least 4 days of maintenance on duloxetine during inpatient admission.
  Number of cocaine doses earned by subjects on a progressive ratio schedule of reinforcement.
Reinforcing Effects of Cocaine Following Methylphenidate Maintenance. | Following at least 4 days of maintenance on duloxetine during inpatient admission.
  Number of cocaine doses earned by subjects on a progressive ratio schedule of reinforcement.
Reinforcing Effects of Cocaine Following Methylphenidate and Duloxetine Maintenance. | Following at least 4 days of maintenance on methylphenidate and duloxetine during inpatient admission.
  Number of cocaine doses earned by subjects on a progressive ratio schedule of reinforcement.

SECONDARY OUTCOMES:
Adjective Rating Scale-Sedative | Nine times over approximately four weeks inpatient admission.
  Subjects will complete the adjective rating scale during nine sessions while they are admitted to our inpatient unit. Responses to 16 items are summed (total score=0-64; Higher values=more sedation) to calculate scores on a sedative subscale.
Adjective Rating Scale-Stimulant | Nine times over approximately four weeks inpatient admission.
  Subjects will complete the adjective rating scale during nine sessions while they are admitted to our inpatient unit. Responses to 16 items are summed (total score=0-64; Higher values=more stimulation) to calculate total scores on a stimulant subscale.
Drug Effect Questionnaire | Nine times over approximately four weeks inpatient admission.
  Subjects will complete the drug effect questionnaire during nine sessions while they are admitted to our inpatient unit. The items (total scores=0-100; Higher scores=greater drug effect) on this scale categorize the constellation of drug effects endorsed by subjects.
Heart rate | Daily over approximately four week inpatient admissions.
  Beats per minute. Measured daily during inpatient admission.
Blood pressure | Daily over approximately four week inpatient admissions.
  mmHg.Measured daily during inpatient admission.
Temperature | Daily over approximately four week inpatient admissions.
  Degrees fahrenheit. Measured daily during inpatient admission.
Side effects | Daily over approximately four week inpatient admissions.
  Subjects will complete a side effects questionnaire daily while they reside on the inpatient unit. Side Effects questions will query subjects about common effects of centrally active medications.
Delay Discounting Task | Nine times over approximately four weeks inpatient admission.
  Subjects will complete the delay discounting task during nine sessions while they are admitted to our inpatient unit. Responses will be used to calculate discounting slope (i.e., K).
Attentional Bias | Nine times over approximately four weeks inpatient admission.
  Subjects will complete attentional bias during nine sessions while they are admitted to our inpatient unit. Time attending to drug stimuli will be used to evaluate attentional bias.
Inhibitory Control | Nine times over approximately four weeks inpatient admission.
  Subjects will complete an inhibitory control task during nine sessions while they are admitted to our inpatient unit. Ability to inhibit prepotent responding will be used to calculate inhibitory control.

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Rush, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No